CLINICAL TRIAL: NCT01445704
Title: Use of Probiotics to Aid in Weight Loss
Acronym: Probiotics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prisma Health-Upstate (Other)
Collaborators: Xymogen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00006473
Record Dates: First submitted 2011-09-29; First posted 2011-10-04 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-04

CONDITIONS: Weight Loss
Keywords: Weight loss; Probiotics; Gastric Bypass
MeSH Terms: conditions — Weight Loss | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotics (Experimental): Patients treated with a probiotic (in capsule form) once daily for 12 weeks
  Interventions: Dietary Supplement: Probiotics
- Placebo (Placebo Comparator): Patients treated with a placebo (in capsule form) identical to that of the probiotic capsule once daily for 12 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotics — The probiotic supplementation will use lactic acid bacteria in the "ProbioMax DF™" supplement from Xymogen, Inc. This preparation consists of a four-strain probiotic with 100 billion CFU per vegetable capsule. The strains included are Lactobacillus acidophilus La-14, Bifidobacterium lactis HN019, Lactobacillus planarum Lp-115, and Bifidobacterium longum B1-05.
  Arms: Probiotics
Dietary Supplement: Placebo — The placebo supplementation is identical-looking to the capsule of the probiotic supplementation.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the success of daily supplementation of multiple probiotic bacterial cultures over 12 weeks in increasing the percentage of excess weight loss in the RNYGB (Gastric Bypass) weight loss population.

DETAILED DESCRIPTION:
Hypothesis:

The daily supplementation of a probiotic will increase weight loss compared to a placebo supplement in the post-operative gastric bypass patients.

Study Design:

All patients in this study will be scheduled to undergo the RNYGB (Gastric Bypass) procedure to assist in weight loss. Patients in this study will be randomized to one of two groups: Group 1 (Probiotics) or Group 2 (Placebo). Patients will begin supplementation at the beginning of their 4 week pre-surgery Optifast© 800 diet. All patients will take supplements for a total of 12 weeks. Nutritional education and support will be provided to each patient enrolled in the study. Weight loss will be measured using a machine that measures body composition. All patients will complete a quality of life questionnaire with regard to gastrointestinal health and a hair loss survey pre treatment and at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female at least 18 years of age
* Signed informed consent
* Willingness to take a supplement once a day for 12 weeks
* Undergoing a RNYGB (gastric bypass) procedure
* Willingness to complete quality of life questionnaire and hair loss survey

Exclusion Criteria:

* Pregnant Female
* Lactating Female
* Male or Female less than 18 years of age
* Patients on chronic antibiotic treatment (prescribed more than 2 courses of antibiotics over the 12 week study period)
* Patients who have demonstrated medical therapy non-compliance past or present

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2010-06; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Percentage of weight loss in post operative gastric bypass patients. | 12 weeks
  Percentage of weight loss will be measured using the The RJL Systems' Quantum IX on all patients for bioelectrical impedance analysis (BIA) to assess human body composition before beginning supplementation and at the end of the 12 week period. The Tanita system will be used as the back-up machine throughout the study as applicable.

SECONDARY OUTCOMES:
Impact of study medication (Probiotics vs. Placebo) on overall Gastrointestinal Health | 12 weeks
  Use of the validated quality of life survey: GIQOLI (Gastrointestinal Quality of Life Index)

CONTACTS AND LOCATIONS:
Overall Officials: John D Scott, M.D., Principal Investigator — Prisma Health-Upstate
Locations (1):
- Greenville Hopsital System - Division of Bariatric and Minimal Access Surgery, Greenville, South Carolina, United States

REFERENCES:
- [Background] Anderson JW, Gilliland SE. Effect of fermented milk (yogurt) containing Lactobacillus acidophilus L1 on serum cholesterol in hypercholesterolemic humans. J Am Coll Nutr. 1999 Feb;18(1):43-50. doi: 10.1080/07315724.1999.10718826. PMID 10067658
- [Background] Vanderhoof JA. Probiotics: future directions. Am J Clin Nutr. 2001 Jun;73(6):1152S-1155S. doi: 10.1093/ajcn/73.6.1152S. PMID 11393194
- [Background] Kopp-Hoolihan L. Prophylactic and therapeutic uses of probiotics: a review. J Am Diet Assoc. 2001 Feb;101(2):229-38; quiz 239-41. doi: 10.1016/S0002-8223(01)00060-8. PMID 11271697
- [Background] Woodard G.; Peraza J.; Downey J.; Encarnacion B.; Morton J. 343 Probiotics Improve Weight Loss, GI-Related Quality of Life and H2 Breath Tests After Gastric Bypass Surgery: A Prospective Randomized Trial. Gastroenterology. 2008 April; Vol. 134 (4), suppl. 1, pp. A-846.
- [Background] Eypasch E, Williams JI, Wood-Dauphinee S, Ure BM, Schmulling C, Neugebauer E, Troidl H. Gastrointestinal Quality of Life Index: development, validation and application of a new instrument. Br J Surg. 1995 Feb;82(2):216-22. doi: 10.1002/bjs.1800820229. PMID 7749697